CLINICAL TRIAL: NCT07055659
Title: Enhancing Oral Hygiene in Children Through an Innovative Motivational Model: A Randomized Controlled Trial
Brief Title: Enhancing Oral Hygiene in Children Through an Innovative Motivational Model
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Wesam Fathi, Assistant Professor of Periodontology, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Qassim University "21-16-15"
Record Dates: First submitted 2025-06-21; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Oral Hygiene Orientation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): group with plant: this is the experimental group: the child will be given a plant to water it during 2-minute brushing habit. DMF, Plaque index and gingival index (describing number of decayed teeth and and status of gingiva with the amount of plaque) all will be compared between the groups at the beginning and at the end of the study.
  Interventions: Diagnostic Test: Oral hygiene assessment
- Group B (Placebo Comparator): group without plant: the control or placebo group: the child will not receive a plant but is instructed to brush his teeth for 2-minutes and keep this brushing habit for the whole period of the study.
  DMF, Plaque index and gingival index (describing number of decayed teeth and and status of gingiva with the amount of plaque) all will be compared between the groups at the beginning and at the end of the study.
  Interventions: Diagnostic Test: Oral hygiene assessment

INTERVENTIONS:
Diagnostic Test: Oral hygiene assessment — experimental group will be given a plant to water it during 2-minute brushing habit. number of decayed teeth and and status of gingiva with the amount of plaque will be compared between the groups
  Other Names: DMF; Plaque Index; Gingival Index

SUMMARY:
Background

Children are susceptible to dental caries and periodontal disease, which are both preventable.

Anxiety and fear of dental pain and dentists are common among children worldwide, so it is important to encourage new strategies to overcome this condition.

Illustrations and visual aids may be helpful in passing along oral hygiene instructions to children.

Rationale As a visual model, watering the plant is linked to brushing time. The evident growth of the plant as monitored by the child, can be helpful to instill the importance of maintaining proper dental hygiene.

Study objectives To motivate children to maintain proper oral health care.

Methods Forty 8 to 12 years old children (20 boys and 20 girls) will be randomly selected. Clinical oral examination is conducted to evaluate the dental caries and oral status gingival status of all children. Parents were asked to answer a simple questionnaire to assess oral health behaviors of their kids.

DETAILED DESCRIPTION:
Introduction Children are susceptible to dental caries and periodontal disease, which are both preventable. (1) Poorly understood dental hygiene behaviors are considered factors that contribute to the prevalence of dental caries and plaque accumulation among children. (2) Moreover, anxiety and fear of dental pain and dentists are common among children worldwide, so it is important to encourage new strategies to overcome this condition. (3) Children's intention to improve oral hygiene behavior can be improved by addressing psychological and behavioral obstacles when creating positive social motivation. (4) Illustrations and visual aids may be helpful in passing along oral hygiene instructions to children. (5) When motivational methods were applied during toothbrushing, e.g. an hourglass timer or a music video, a statistically significant decrease was observed in Plaque Index and Gingival Index values. (6) In light of oral health contributes significantly to the promotion of general health and the prevention of chronic diseases. (7) As a result, both oral disease prevention and oral health promotion should be incorporated into chronic disease prevention and health promotion programs. (8) As a visual model, watering the plant is linked to brushing time. The evident growth of the plant as monitored by the child, can be helpful to instill the importance of maintaining proper dental hygiene.

3. Research objectives The study aims to motivate children to maintain proper oral health care. Materials and methods Prospective, randomized, clinical trial study. 4.2.Study setting: Dental clinics at, college of dentistry, Qassim University 4.3.Study duration: three years. The study is estimated to be three years. 4.4.Sample size: The sample size are forty children between 8-12 years old 4.5.Sampling technique (with inclusion and exclusion criteria): Forty children will be randomly selected from the dental clinics of Qassim University. 40 medically -free children (20 boys and 20 girls) of age 8-12 years old are involved in the study. Any child with any physical or mental disability will be excluded. Moreover, puberty is a reason for exclusion too. The collected sample will be equally divided, into four groups with equal gender distribution. For boys ( Group A AND Group B),For girls ( Group A AND Group B).

Study sample: Group A Experimental sample: Group B Each group (A+B) will be given a toothbrush and toothpaste, and the explain to them correct oral hygiene..

For group B we will given him also the plant as a motivation . 4.6.Data collection methods:

1. Clinical examination: the following clinical parameters are recorded: DMF and df, Gingival index, and Plaque index, using periodontal probe, dental explorer. Data will be collected on the first and last visit ( in day zero and day 90)
2. Questionnaire: to assess oral health behaviors of the kids will be in the last visit (in day 90) for the parent 4.8.Data management and analysis plan: The collected data will be kept at the College of Dentistry - Qassim University No data access will be granted to unauthorized individuals. The data will be analyzed statistically. The descriptive data related to caries and plaque accumulation will be descriptively analyzed. The parent was asked to answer questionnaire for assessed on their oral health behaviors. The children age and gender will be calculated. Caries, gingival and plaque indices are used to assess plaque accumulation and evaluate the condition of the teeth and the gingiva. The questionnaire collected data would assess the of the child's interest in home care. The collected parameters will be collected and recorded in an Excel sheet and statistically analyzed. Data will be collected at baseline and after three months and will be analyzed using Statistical Package for Social Sciences (SPSS) version 21.0 .

4.9.Ethical considerations: The nature of the study will be explained to the mother of the child and informed consent will be obtained. No access will be granted to the code key to any unauthorized individuals.

ELIGIBILITY:
Inclusion Criteria:

* medically -free children

Exclusion Criteria:

* Any child with any physical or mental disability will be excluded. puberty is a reason for exclusion too

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical examination: Oral hygiene status | 90 days
  the following clinical parameters are recorded: DMF and df, Gingival index, and Plaque index, using periodontal probe, dental explorer. Data will be collected on the first and last visit ( in day zero and day 90).
  DMF and df are expressed in number of decayed, missed or filled teeth at the beginning and at the end of the study. any increase would express worse situation.
  Gingival index expresses inflammation in gingiva, that happens when gingiva is diseased (due to poor oral hygiene). the scores are 0-3, the higher the worse the situation.
  Plaque index represents the amount of accumulated plaque, scored 0-3, the higher the worse the situation.
  all records are taken at the beginning and at the end of the study, to compare the effect of giving a plant to the explementary group would or wouldn't improve oral hygiene of the child (less plaque) and preserve gingival health (less gingival index) and teeth (less DMF changes).

SECONDARY OUTCOMES:
Questionnaire | 90 days
  to assess oral health behaviors of the kids will be in the last visit (in day 90) for the parent.
  The following questions are to be answered by parents:
  Did your child show interest when watering his plant? Does your child brush himself twice a day? Does your child continue to water his plant twice a day? Did the growth of the plant motivate your child to continue brushing his teeth Do you think that your child's care for plants has encouraged him and increased his interest in oral health?
  the answers are only yes or no to describe child's commitment to oral hygiene

CONTACTS AND LOCATIONS:
Locations (1):
- Qassim University, Buraidah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
gender and age
Supporting Information: Study Protocol